CLINICAL TRIAL: NCT03074396
Title: Usefulness of a Mobile Information Management System for Haemodialysis Patients and the Prospect of Participatory Medicine
Brief Title: Usefulness of a Mobile Information Management System for Haemodialysis Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Hoseok Koo, Assistant professor, Inje University Seoul Paik Hospital, Inje University
Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: DialysisNet
Record Dates: First submitted 2017-02-25; First posted 2017-03-08 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Quality of Life; Drug Habit
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- before and after use of program (Other): one arm (10 patients and 4 physicians) before and after use of dialysisNet (for doctors) and Avatar Beans (for patients)
  Interventions: Device: Use of DialysisNet for doctor; Device: Use of Avatar Beans for patient

INTERVENTIONS:
Device: Use of DialysisNet for doctor — DialysisNet is mobile application for physicians for haemodialysis patients. Patient-centred data integration and exchange were based on the American Society for Testing and Materials Continuity of Care Record standard.
Device: Use of Avatar Beans for patient — Avatar Beans is mobile application for haemodialysis patients. Patient-centred data integration and exchange were based on the American Society for Testing and Materials Continuity of Care Record.

SUMMARY:
The investigators developed and used the DialysisNet mobile application for physicians and Avatar Beans mobile application for haemodialysis patients. Patient-centred data integration and exchange were based on the American Society for Testing and Materials Continuity of Care Record standard. The investigators enrolled 10 patients and 4 physicians. Questionnaires to evaluate user experience and usefulness were administered before and after use.

ELIGIBILITY:
Inclusion Criteria:

* patients who have maintenance hemodialysis treatment
* accept consent form

Exclusion Criteria:

* pregnant

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The change of Short Form 36 questionnaire for quality of life | 3 month after the use of DialysisNet (for doctors) and Avatar Beans (for patients)

SECONDARY OUTCOMES:
The change of morisky medication adherence scale (MMAS) for drug compliance | 3 month Before and after the use of DialysisNet (for doctors) and Avatar Beans (for patients)

IPD SHARING:
Plan to Share IPD: No